CLINICAL TRIAL: NCT01593670
Title: Decitabine and Vorinostat With CD3/CD19 Depleted Haploidentical Donor Natural Killer (NK) Cells for the Treatment of High Risk Myelodysplastic Syndromes (MDS)
Brief Title: Decitabine and Vorinostat Conditioning Followed by CD3-/CD19- NK Cells Infusion for High Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011LS124; MT2012-04 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Myelodysplastic Syndrome
Keywords: high risk myelodysplastic syndrome; natural killer cells
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; Vorinostat; Interleukin-2; Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients With High Risk MDS (Experimental): Patients who received treatment for high risk myelodysplastic syndromes (MDS). Treatment Received: Decitabine 10 mg/m^2/day intravenous (IV) over 1 hour days 1-5; Vorinostat 200 mg by mouth (PO) twice a day days 6-15; Il-2 activated donor natural killer cells (NK) infusion IV over 15 to 60 minutes day 17; Interleukin-2 6 million units subcutaneous (SQ) 3 times a week for 3 doses beginning day 17. Repeat treatment course 6 to 8 weeks after cycle 1 start date.
  Interventions: Drug: Decitabine; Drug: Vorinostat; Biological: Interleukin-2; Other: Natural killer (NK) cells

INTERVENTIONS:
Drug: Decitabine — administered intravenous (IV), 10 mg/m^2/day over 1 hour on days 1-5.
  Other Names: Dacogen
Drug: Vorinostat — 200 mg by mouth (PO) twice a day on days 6-15
  Other Names: Zolinza
Biological: Interleukin-2 — 6 million Units subcutaneous (SQ) 3 times a week for 3 doses beginning day 17
  Other Names: IL-2
Other: Natural killer (NK) cells — infusion intravenously (IV) over 15 to 60 minutes day 17

SUMMARY:
This is a Phase II therapeutic trial combining Decitabine days 1-5 with oral Vorinostat twice daily days 6-15 followed by a single infusion of CD3-/CD19- enriched donor natural killer (NK) cells on day 17 and a short course of Interleukin-2 (IL-2) to facilitate NK cell survival and expansion. Two courses of treatment will be given separated by 6-8 weeks. The intent is to administer all treatment in the outpatient setting.

DETAILED DESCRIPTION:
A single donor apheresis will be collected on day 15 of cycle 1, enriched for NK cells with the large scale CliniMacs device (Miltenyi) and activated by overnight incubation with IL-2. After washing, the final NK cell product will be divided in two, with half given fresh on day 17 of course #1 and half stored frozen until day 17 of course #2.

Clinical response will be formally assessed 4-6 weeks after the start of 2nd course based on International Working Group (IWG) criteria; however, bone marrow evaluations will be completed to assess for any sign of significant disease progression between cycle 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high risk myelodysplastic (MDS) that meets one of the following disease classifications and is requiring treatment:

  * International Prognostic Scoring System (IPSS) Category: INT-2 or High Risk
  * WHO Classification: RAEB-1 or RAEB-2
  * High risk cytogenetic abnormality as defined by presence of Monosomy 7, complex karytope, or monosomal karyotype
  * WHO Based Prognostic Scoring System (WPSS): High or Very High Risk
* Patients may be untreated or have had a maximum of 2 cycles of hypomethylating agents (azacitidine or decitabine) without evidence of treatment failure as defined by progression to more advanced MDS Who classification or AML. Patients must not have received treatment for their MDS within 4 weeks of beginning the trial. Treatments allowed prior to that time include azacitidine or decitabine and hematopoietic growth factors. No prior AML-like induction therapy allowed.
* Age ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Available related HLA-haploidentical NK cell donor by at least Class I serologic typing at the A&B locus
* Have acceptable organ function within 14 days of enrollment
* Ability to be off prednisone and other immunosuppressive drugs for at least 3 days prior to the natural killer (NK) cell infusion
* Women of child bearing potential must agree to use effective methods of contraception
* Voluntary written consent

Exclusion Criteria:

* Pregnant or lactating.
* Prior 7 + 3 (cytarabine given continuously for 7 days with an anthracycline drug, such as daunorubicin or idarubicin given for the 1st 3 days of treatment) or other AML-type induction chemotherapy
* New progressive pulmonary infiltrates on screening chest x-ray or chest computed tomography (CT) scan that has not been evaluated with bronchoscopy (when feasible)
* Uncontrolled bacterial or viral infections - chronic asymptomatic viral hepatitis is allowed
* Pleural effusion moderate to large in size that are detectable on chest xray
* Known hypersensitivity to one or more of the study agents
* Prior hypomethylating treatment greater than 2 cycles or with documented treatment failure
* Prior use of histone deacetylase inhibitors
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study in the opinion of the enrolling investigator
* Inability to swallow capsules
* Active human immunodeficiency virus (HIV)
* Other active and potentially life threatening malignancy excluding localized basal or squamous cell skin cancer, cervical carcinoma in situ, superficial bladder cancer, localized prostate cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Warlick, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With High Risk MDS
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With High Risk MDS
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Achieved a Clinical Response
Description: Clinical response includes: Complete Response (less than 5% myeloblasts present in the bone marrow and in the peripheral blood a hemoglobin of at least 11g/dl, platelets of at least 100 X 10E9/L, neutrophils of at least 1.0 X 10E9/L, and blasts 0%); Partial Response (all Complete Response criteria if previously abnormal except bone marrow myeloblasts are decreased by more than 50% over pre-treatment, but still greater than 5%); and hematologic improvement (a hemoglobin increase of greater than 1.5g/dl or decreased red blood cell transfusions by at least 4 per 8 week period, a platelet increase of more than 30 X 10E9/L for patients with a baseline of more than 20 X 10E9/L or an increase by 100% for those with a baseline of less than 20 X 10E9/L, and a neutrophil increase of at least 100% and an absolute increase of greater than 0.5 X 10E9/L.
Time Frame: After 2 Courses of Treatment (Approx. 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With High Risk MDS
Number analyzed (Participants) | 9
Participants | 5

2. Secondary Outcome: Number of Patients Who Experienced Grade 3 or Higher Non-hematologic Adverse Events
Description: Adverse events (AEs) will be graded using Common Terminology Criteria for Adverse Events v4.0 (CTCAE). Non-hematologic adverse events are defined as untoward medical occurrences associated with the use of a study drug whether or not considered study drug related, excluding those events involving white blood cells, neutrophils, red blood cells or platelets. In general, grade 3 AEs are defined as 1) being severe or medically significant but,not immediately life-threatening; 2) requiring hospitalization or prolongation of hospitalization; 3) disabling; or 4) limiting self care activities. Grade 4 AEs are defined as 1) having life-threatening consequences; or 2) requiring urgent intervention. Grade 5 AEs are defined as causing death related to an adverse event.
Time Frame: Day 1 through Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With High Risk MDS
Number analyzed (Participants) | 9
Participants | 7

3. Secondary Outcome: Number of Patients Who Became Transfusion Independent
Time Frame: 4-6 Months Post Start of Cycle 1
Population: 7 of the 9 patients were not evaluable for this outcome measure - 5 went on to stem cell transplant and 2 died before reaching the 4-6 month post start of cycle 1 milestone.This left 2 evaluable patients for the outcome measure, and thus this endpoint is not informative due to lack of evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With High Risk MDS
Number analyzed (Participants) | 2
Participants | 0

4. Secondary Outcome: Number of Patients Who Had Natural Killer (NK) Cell Expansion
Description: NK cell expansion is defined as the presence of donor NK cells in the recipient at Day 8 post NK cell infusion.
Time Frame: After Cycle 2 (approx. 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With High Risk MDS
Number analyzed (Participants) | 9
Participants | 0

5. Secondary Outcome: Overall Survival
Description: Patients alive at 1 year.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With High Risk MDS
Number analyzed (Participants) | 9
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Patients With High Risk MDS
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With High Risk MDS (N=9)
Hypotension (Vascular disorders) | 1
Renal Colic (Renal and urinary disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Otomastoiditis (Ear and labyrinth disorders) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1
Infection, Source Unknown (Infections and infestations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With High Risk MDS (N=9)
Chills (General disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine Increased (Investigations) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Edema, NOS (General disorders) | 4
Fatigue (General disorders) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 6
Fever (General disorders) | 4
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Infusion Related Reaction (General disorders) | 2
Injection Site Reaction (General disorders) | 6
Itchy Nose (Skin and subcutaneous tissue disorders) | 1
Nasal Drainage (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Para-Influenza (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
White Blood Cell Decreased (Investigations) | 4
Neutrophil Count Decreased (Investigations) | 7
Platelet Count Decreased (Investigations) | 7
Bacteremia (Infections and infestations) | 1
Cellulitis, Toe (Infections and infestations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Blood Bilirubin Increased (Investigations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholesterol High (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 2
Ear Pain (Ear and labyrinth disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Edema, Ankle (General disorders) | 1
Pain, Toe (Musculoskeletal and connective tissue disorders) | 1
Renal Calculi (Renal and urinary disorders) | 1
Renal Colic (Renal and urinary disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT01593670/Prot_SAP_000.pdf